CLINICAL TRIAL: NCT04744363
Title: Phase 1, FIH, Randomized, Double-blind, Single-dose, Parallel-group, 3-arm Study Comparing the PK, Safety, Tolerability, and Immunogenicity Profiles of AVT04, EU-approved Stelara®, and US-licensed Stelara® in Healthy Adult Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability Study of AVT04 to EU Approved and US Licensed Stelara (Ustekinumab)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVT04-GL-101
Record Dates: First submitted 2020-12-16; First posted 2021-02-09 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Intervention Model Description: A Phase 1, first-in-human, randomized, double-blind, single-dose, parallel-group, 3-arm study comparing the pharmacokinetic, safety, tolerability, and immunogenicity profiles of AVT04, EU approved Stelara®, and US licensed Stelara® in healthy adult subjects
Who Masked: Investigator
Masking Description: Blinded and unblinded site teams
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AVT04 45 mg SC (Experimental): Single dose Pre-filled syringe to be injected subcutaneously into thigh or abdomen
  Interventions: Drug: Stelara PFS
- US Stelara 45 mg SC (Active Comparator): Single dose Pre-filled syringe to be injected subcutaneously into thigh or abdomen
  Interventions: Drug: Stelara PFS
- EU Stelara 45 mg SC (Active Comparator): Single dose Pre-filled syringe to be injected subcutaneously into thigh or abdomen
  Interventions: Drug: Stelara PFS

INTERVENTIONS:
Drug: Stelara PFS — Pre filled syringes filled with AVT04 and Stelara
  Other Names: Ustekinumab

SUMMARY:
Protocol Title:

A Phase 1, first-in-human, randomized, double-blind, single-dose, parallel-group, 3-arm study comparing the pharmacokinetic, safety, tolerability, and immunogenicity profiles of AVT04, EU approved Stelara®, and US-licensed Stelara® in healthy adult subjects

Short Title:

A first-in-human randomized, double-blind study to compare AVT04 with EU-approved Stelara and US-licensed Stelara as a single-dose subcutaneous injection in healthy adult subjects

Rationale:

Alvotech (hereafter, the Sponsor) is developing AVT04 globally as a proposed biosimilar to the reference product Stelara (ustekinumab) for subcutaneous (SC) use. This is a first-in-human (FIH) clinical study with AVT04. The study aims to demonstrate pharmacokinetic (PK) similarity of the proposed biosimilar test product AVT04 and the reference products EU approved Stelara and US-licensed Stelara, in addition to evaluating the safety and tolerability of AVT04, when administered as a single 45 mg/0.5 mL SC dose.

DETAILED DESCRIPTION:
Overall Design:

This study is designed as a FIH, multicenter, randomized, double-blind, 3-arm, parallel-group study of AVT04 compared with EU-approved and US-licensed Stelara when administered as a single 45 mg/0.5 mL SC injection in healthy adult subjects.

Subjects will undertake a Screening visit between Day -28 and Day -1 to determine their eligibility in the study. Subjects who meet the eligibility criteria will be admitted to the study site on the day prior to dosing (Day -1), during which their continued eligibility will be assessed up to Day 1 prior to dosing. On Day 1, eligible subjects will be randomized and will receive a single dose of one of the following: AVT04, US licensed Stelara, or EU approved Stelara.

A staggered sentinel dosing strategy will be implemented as a safety measure, with equal numbers of subjects randomized to each treatment: Sentinel Group 1 (n = 3 subjects [1 per group]), Sentinel Group 2 (n = 6 subjects [2 per group]), and Sentinel Group 3 (n = 9 subjects [3 per group]). Following investigational product (IP) administration, there will be at least 72 hours of close observation and safety monitoring by the Principal Investigator (PI) for each subject and between sentinel groups (ie, 72 hours should have elapsed following IP administration for the last subject in each sentinel group). Provided there are no significant safety or tolerability concerns (or events that meet the study stopping criteria) in the previous sentinel group following a safety review and discussion between the PI, Medical Monitor, and Sponsor, the next sentinel group of subjects will be randomized and dosed. Once the IP dose is deemed to be safe and well tolerated in all 3 sentinel groups, the remaining subjects (n = 276 subjects [92 subjects per group]) will be randomized and dosed.

Sentinel subjects will remain confined to the study site from Day -1 to Day 4 (72 hours postdose); all remaining subjects will be confined to the study site from Day -1 up to Day 2 (24 hours postdose). Following dosing, PK, safety, tolerability, and other assessments will be performed according to the Schedule of Assessments. Subjects will return to the study site on an outpatient basis daily up to Day 12, then once a week from Day 15 to Day 64, followed by once every 2 weeks up to Day 78, and finally on Day 92 for the End-of-Study (EOS) visit.

Number of Subjects:

Approximately 294 healthy subjects (98 per group) are planned to be enrolled at multiple study sites in New Zealand and Australia. Efforts will be made to include at least 10% of subjects (30 subjects, approximately 10 per group) who are of Japanese origin or ethnicity (defined as a second-generation Japanese person living abroad or born in Japan; and both parents and grandparents are of Japanese origin).

A total of 45 subjects (15 per group) are planned to be included in the exploratory ex-vivo biomarker sub study.

Treatment Groups and Duration:

Eligible subjects will be randomly assigned in a 1:1:1 ratio to receive a single 45 mg/0.5 mL SC dose of ustekinumab as AVT04 (test product) or US licensed Stelara or EU approved Stelara (reference products) on Day 1. Randomization will be stratified by ethnicity and body weight at Day -1 as follows: Japanese, non Japanese ≤80 kg, and non-Japanese >80 kg.

The study duration per subject will be approximately 17 weeks. The study will consist of a 4 week Screening period, a 13-week treatment period and assessment period, and an EOS visit on Day 92.

Study Stopping Criteria:

If either of the following scenarios occur, study enrollment and dosing will be halted:

* If >2 subjects experience a suspected unexpected serious adverse reaction (defined as an adverse event [AE] that is serious, unexpected, and considered related to the IP).
* If the Sponsor or Investigator considers there to be an unfavorable benefit-risk ratio based on emerging safety data.

If following consultation between the PI, Medical Monitor, and Sponsor, it is considered appropriate to restart study drug administration in the remaining subjects, justification will be submitted to the Health and Disability Ethics Committee/Human Research Ethics Committee for restarting the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all of the following criteria apply at any time starting from Screening up to Day 1 prior to IP administration:

1. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol.
2. Male or female subjects.
3. Subjects must be 18 to 55 years old inclusive, at the time of signing the ICF.
4. Have a body weight of 60.0 to 90.0 kg (inclusive) and body mass index (BMI) of 18.5 to 30.0 kg/m2 (inclusive).
5. For Japanese subjects only Is a second-generation Japanese person living abroad and both parents and grandparents are of Japanese origin, OR Was born in Japan and both parents and grandparents are of Japanese origin.
6. Medical history without major pathology, according to the PI's judgment.
7. Resting supine systolic blood pressure (BP) of ≤140 mm Hg and diastolic BP of ≤90 mm Hg; other vital signs showing no clinically relevant deviations according to the PI's judgment.
8. Computerized (12-lead) electrocardiogram (ECG) recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the PI.
9. Glycated hemoglobin (HbA1c) ≤42 mmol/mol.
10. Clinical safety laboratory results are within the reference ranges or showing no clinically relevant deviations as judged by the PI.
11. Have a negative urine drug screen (opiates, methadone, cocaine, amphetamines [including ecstasy and methamphetamines], cannabinoids, barbiturates, and benzodiazepines) and a negative alcohol breath test.
12. Tested negative for TB, hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (anti-HBc), anti-hepatitis C virus (HCV) antibodies, and anti-human immunodeficiency virus (HIV) 1/2 antibodies at Screening.
13. Nonsmoker or occasional smoker, ie, smokes ≤10 cigarettes (or equivalent of tobacco- or nicotine containing products) per week within 3 months of Screening, and ability and willingness to refrain from smoking during confinement at the study site.
14. Ability and willingness to abstain from alcohol from 48 hours prior to drug administration, during confinement at the study site until discharge, and 24 hours prior to ambulatory visits.
15. Female subjects are eligible to participate if they are not pregnant (see Appendix 3), not breastfeeding, and at least ONE of the following conditions applies:

    1. Is not a woman of childbearing potential (WOCBP), defined as:

       Surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, as confirmed by review of the subject's medical records, medical examination, or medical history interview), or Postmenopausal (defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone [FSH] level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy [HRT]. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient). Female subjects on HRT and whose menopausal status is in doubt will be required to use 1 of the non estrogen hormonal highly effective contraception methods (Appendix 3) from Screening (signing the ICF) until at least 13 weeks after IP administration if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.
    2. Is a WOCBP who agrees to use a highly effective method of contraception (Appendix 3) consistently and correctly from Screening (signing the ICF) until at least 13 weeks after IP administration.
16. Nonsterilized male subjects with female partners of childbearing potential are eligible to participate if they agree to ONE of the following from Screening (signing the ICF) until at least 13 weeks after IP administration:

    1. Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.
    2. Agree to use a male condom and have their partner use of a contraceptive method with a failure rate of <1% per year as described in Appendix 3 when having penile-vaginal intercourse with a WOCBP who is not currently pregnant.
    3. Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse or use a male condom during each episode of penile penetration.
17. In addition, male subjects must refrain from donating sperm from Screening (signing the ICF) until at least 13 weeks after IP administration.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply at any time starting from Screening up to Day 1 prior to IP administration:

1. Have a history of relevant drug and/or food allergies.
2. Have a history of hypersensitivity to Stelara, AVT04, or their constituents.
3. Have a known history of previous exposure to IL-12 and/or IL-23 inhibitors.
4. Have any past or concurrent medical conditions that could potentially increase the subject's risks or that would interfere with the study evaluation, procedures, or study completion. Examples of these include medical history with evidence of clinically relevant pathology (eg, malignancies or demyelinating disorders).
5. Presence of chronic obstructive pulmonary disease. Childhood asthma is allowed.
6. Presence of type 1 or 2 diabetes mellitus.
7. Have a known history of active or latent TB, except for subjects with documented and complete adequate treatment of TB or initiation (>1 month) of adequate prophylaxis of latent TB, with an isoniazid-based regimen.
8. Have resided or traveled in regions where tuberculosis and mycosis are endemic within 90 days before Screening, or who intend to visit such a region during the study period or within 3 months (12 weeks) after dosing.
9. Any current active infections, including localized infections, or any recent history (within 1 week prior to study drug administration) of active infections (including severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] based on a positive COVID-19 polymerase chain reaction [PCR] nasopharyngeal swab test), cough or fever, or a history of recurrent or chronic infections.
10. Participation in a clinical study with an IP within 60 days or 5 half-lives of that IP (if known), whichever is longer, prior to IP administration in the current study.
11. Treatment with nontopical medications (including over-the-counter [OTC] medications and herbal remedies such as St. John's Wort extract) within 7 days or 5 half lives of the drug (whichever is longer) prior to IP administration, with the exception of multivitamins, vitamin C, food supplements and a limited amount of acetaminophen (up to 2 g in 24 hours, but <1 g in 4 hours) or ibuprofen (<1.2 g per day), which may be used throughout the study.
12. Have received live vaccines during the past 4 weeks before Screening or have the intention to receive vaccination during the study period or within 13 weeks after dosing.
13. Donation of more than 500 mL of blood within 8 weeks prior to drug administration.
14. History of alcohol abuse (with an average intake exceeding 10 drinks/week for women and 15 drinks/week for men: 1 drink = 360 mL of beer, 150 mL of wine, or 45 mL of spirits) or drug addiction (including soft drugs like cannabis products).
15. Any persons who are:

    1. An employee of the study site, Investigator, contract research organization (CRO) or Sponsor;
    2. A first-degree relative of an employee of the study site, the Investigator, CRO, or the Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 294 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-03-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve AUC0-inf | From Baseline to day 92
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUC 0-t) of AVT04, US Stelara EU Stelara
Maximum serum concentration | From Baseline to day 92
  Venous blood samples will be collected for measurement of serum concentration of AVT04, EU Stelara, US Stelara

SECONDARY OUTCOMES:
Ustekinumab serum concentration-time profile following single-dose administration | From Baseline to day 92
  Venous blood samples will be collected for measurement of serum concentration time profile of AVT04, US-Stelara EU Stelara
The secondary PK parameters to be assessed are: AUC0-t | From Baseline to day 92
  Venous blood samples will be collected for measurement of the title measures of AVT04, US-Stelara EU Stelara
Adverse Events | From screening to day 92
  The safety parameters to be assessed include AEs, clinical laboratory assessments (hematology, clinical chemistry, coagulation, urinalysis and urine microscopy), vital signs, ECG, physical examination findings, and injection site reactions
Immunogenicity assessments include ADAs and NAbs | From screening to day 92
  Formation of neutralizing antibodies measured through a validated system
The secondary PK parameters to be assessed are: Tmax | From screening to day 92
  Venous blood samples will be collected for measurement of the title measures of AVT04, US-Stelara EU Stelara
The secondary PK parameters to be assessed are: Kel | From Screening to day 92
  Venous blood samples will be collected for measurement of the title measures of AVT04, US-Stelara EU Stelara
The secondary PK parameters to be assessed are: t1/2 | From Screening to day 92
  Venous blood samples will be collected for measurement of the title measures of AVT04, US-Stelara EU Stelara
The secondary PK parameters to be assessed are: Vz/F | From screening to day 92
  Venous blood samples will be collected for measurement of the title measures of AVT04, US-Stelara EU Stelara
The secondary PK parameters to be assessed are: CL/F | From Screening to day 92
  Venous blood samples will be collected for measurement of the title measures of AVT04, US-Stelara EU Stelara

OTHER OUTCOMES:
The inflammatory cytokine biomarkers to be assessed include: IFN-γ, IL-22, IL-17, IL-5, IL-13, and IL-10 | From screening to day 92
  Venous blood samples will be collected to assess the cytokine biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Paul Duijzings, MSc, Study Director — Program Lead
Locations (4):
- Australia (2):
  - Nucleus Network, Brisbane
  - Nucleus Network Melbourne, Melbourne
- New Zealand (2):
  - ACS, Auckland
  - CCST, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wynne C, Hamilton P, McLendon K, Stroissnig H, Smith M, Duijzings P, Ruffieux R, Otto H, Sattar A, Haliduola HN, Leutz S, Berti F. A randomized, double-blind, 3-arm, parallel study assessing the pharmacokinetics, safety, tolerability and immunogenicity of AVT04, an ustekinumab candidate biosimilar, in healthy adults. Expert Opin Investig Drugs. 2023 May;32(5):417-427. doi: 10.1080/13543784.2023.2215426. Epub 2023 May 23. PMID 37212315